CLINICAL TRIAL: NCT04720781
Title: The Need of Revisiting to an Outpatient Clinic After the Prescription of Vonoprazan or Esomeprazole for 4weeks for Erosive Esophagitis Without Any Appointments
Brief Title: The Need of Revisiting to an Outpatient Clinic After the Prescription of Vonoprazan or Esomeprazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Revisiting
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan (Active Comparator): Vonoprazan (20mg/day) is prescribed for patients with erosive esophagitis
  Interventions: Drug: Vonoprazan
- Esomeprazole (Placebo Comparator): Esomeprazole (20mg/day) is prescribed for patients with erosive esophagitis
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan (20mg/day) is prescribed for 4 weeks.
  Other Names: Esomeprazole
  Arms: Vonoprazan
Drug: Esomeprazole — esomeprazole (20mg/day)
  Arms: Esomeprazole

SUMMARY:
After vonoprazan (20mg/day) or esomeprazole (20mg/day) for 4weeks is prescribed for patients with erosive esophagitis diagnosed by esophagogastroduodenoscopy, the number of patients who will visit our outpatient clinic again due to some reasons without any appointments is compared with vonoprazan group and esomeprazole.

DETAILED DESCRIPTION:
1. Patients who have erosive esophagitis diagnosed by esophagogastroduodenoscopy is enrolled.
2. Vonoprazan (20mg/day) or esomeprazole (20mg/day) is prescribed for 4weeks the patients randomly without next appointments.
3. Some patients may visit our outpatient clinic again due to some reasons without any appointments.
4. The number of the patients who revisit our outpatient clinic again is compared with vonoprazan group and esomeprazole.

ELIGIBILITY:
Inclusion Criteria:

* outpatients belonging to American Society of Anesthesiologists class I or II
* patients have erosive esophagitis diagnosed by esophagogastroduodenoscopy shortly before the prescription

Exclusion Criteria:

* other acid blockers are taken

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The number of patients who revisit our outpatient clinic after the prescription without any appointments | 3 months
  The need to revisit our outpatient clinic again without any appointments may show the patients' satisfaction or dissatisfaction after the prescription of vonoprazan or esomeprazole. The difference in the number between the two groups may show the difference in the effectiveness between the two medicines.

SECONDARY OUTCOMES:
Change of the main symptom with patients after/before medication when the patients revisit again | 3 months
  The ratio of the degree of the main symptom after/before taking the medicine Good 0%- Bad 100%

OTHER OUTCOMES:
Questionnaire on satisfaction with taking the medicine at revisiting | 3months
  The patient's satisfaction is assessed using visual analogue scale (Exellent 100% to very bad 0%).

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No